CLINICAL TRIAL: NCT04211896
Title: The Efficacy and Safety of Anlotinib Combined With Nivolumab as a Second-Line Treatment in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Anlotinib Combined With Nivolumab for Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANPD1-001
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib; Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anlotinib plus nivolumab (Experimental)
  Interventions: Drug: Anlotinib; Drug: Nivolumab

INTERVENTIONS:
Drug: Anlotinib — Anlotinib will be given at a dose of 12mg once daily on days 1-14 of a 21-day cycle.
Drug: Nivolumab — Nivolumab will be given at a dose of 240 mg every 2 weeks (Odd Cycles: Days 1 and 15 and Even Cycles Day 8) per 21 day Cycle.

SUMMARY:
This study evaluates the safety and efficacy of anlotinib in combination with nivilumab as second-line treatment in advanced NSCLC patients. The primary endpoint of the study is progression-free survival (PFS);the secondary endpoints are disease control rate (DCR), objective response rate (ORR), overall survival (OS) and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-75 years old;
2. ECOG PS：0-1,Expected Survival Time: Over 3 months;
3. Subjects with histologically or cytologically confirmed locally advanced and/or advanced NSCLC, with measurable nidus(using RECIST 1.1);
4. For local advanced or advanced NSCLC, disease progression occurred after first-line systemic treatment previously;
5. The negative patients in EGFR&ALK can participate or who positive in EGFR&ALK, have or have not drug tolerance after the treatment with relative targeted drugs;
6. main organs function is normal;
7. Signed and dated informed consent.

Exclusion Criteria:

1. have used Anlotinib before;
2. Small Cell Lung Cancer (including small cell cancer and other kinds of cancer mixed with non-small cell cancer);
3. examined as positive in EGFR&ALK mutation detection and never take the treatment of TKIs;
4. Previously (within 5 years) or presently suffering from other malignancies;
5. Symptomatic or uncontrolled brain metastases;
6. Unstable systemic disease, including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction within 6 months or serious cardiac arrhythmia requiring medication;
7. Pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 6 months
  PFS is defined as the time from the date of treatment to the first date of disease progression or death from any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD (up to 12 months)
  Treatment response are defined as complete response (CR), partial response (PR), stable disease (SD) and progression disease (PD) according to Response Evaluation Criteria in Solid Tumor (RECISIT criteria, version 1.1). The percentage of patients who achieved CR and PR was defined as objective response rate (ORR)
Disease control rate (DCR) | each 42 days up to intolerance the toxicity or PD (up to 12 months)
  Treatment response are defined as complete response (CR), partial response (PR), stable disease (SD) and progression disease (PD) according to Response Evaluation Criteria in Solid Tumor (RECISIT criteria, version 1.1) and the percentage of patients who achieved CR, PR and SD was defined as disease control rate (DCR).
Overall Survival (OS) | 12 months
  OS is calculated from diagnosis to death or last follow-up time.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Until 30 day safety follow-up visit